CLINICAL TRIAL: NCT03296423
Title: A Randomized Clinical Trial for Enhanced Trained Immune Responses Through Bacillus Calmette-guérin Vaccination to Prevent Infections of the Elderly
Brief Title: Bacillus Calmette-guérin Vaccination to Prevent Infections of the Elderly
Acronym: ACTIVATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTIVATE
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Infection; Hospitalization; Mortality
Keywords: BCG vaccination
MeSH Terms: conditions — Infections | interventions — Vaccination; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients vaccinated with placebo or BCG
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): One intradermal injection of 0.1ml of sodium chloride 0.9%
  Interventions: Biological: Placebo
- Vaccination (Active Comparator): One intradermal injection of 0.1ml of BCG (BCG vaccine Bulgaria strain 1331; Intervax)
  Interventions: Biological: Vaccination

INTERVENTIONS:
Biological: Vaccination — Patients discharged from hospital will be vaccinated with one intradermal injection of 0.1ml of BCG vaccine
  Other Names: BCG; Intervax
  Arms: Vaccination
Biological: Placebo — Patients discharged from hospital will be vaccinated with one intradermal injection of 0.1ml of sodium chloride 0.9%
  Other Names: Saline
  Arms: Placebo

SUMMARY:
One small recent trial in elderly volunteers showed that BCG vaccination can protect against infectious complications, while several studies have demonstrated an increased capacity of innate immune responses to react against pathogens. This process, also called trained immunity, generates the hypothesis that BCG vaccination can prevent or delay new infections in the elderly patients and is studied in the ACTIVATE trial

DETAILED DESCRIPTION:
In an era of antimicrobial resistance, where the already existing antimicrobials are not sufficient, the development of new strategies for the prevention and treatment of infections is of great interest. This approach becomes more and more mandatory in our current era of the financial crisis where bacterial infections by multidrug-resistant emerge and impose heavily on the financial burden of the disease. These infections occur more frequently among elderly patients leading to prolonged hospitalization where unfavorable outcome is not infrequent1. Vaccination is the traditional approach of infection prevention. A classic example focusing on the need to prevent morbid re-infection is vaccination with pneumococcal vaccine the incidence of pneumococcal pneumonia and bacteremia is enormously increasing among the elderly2. The principle of vaccination is to develop memory B-lymphocytes so that early and adequate antibody titers are produced upon re-exposure to the same antigen. This is called the memory function of the adaptive immune system.

Well before adaptive immunity develops proper recognition of a bacterial pathogen is done through binding of well-preserved structures known as pathogen-associated molecular patterns (PAMPs) on pattern-recognition receptors (PRRs) of the innate immune system and mainly of blood monocytes and tissue macrophages. Through a series of experiments in cell systems and animals, it was found that exposure of macrophages to small amounts of PAMPs like the β-glucan of Candida albicans and constituents of Mycobacterium tuberculosis may prevent death upon re-exposure to lethal bacterial challenges like C.albicans and Staphylococcus aureus3-6. Initial exposure to small amounts of PAMPs leads to epigenetic changes that induce the capacity of macrophages and monocytes to produce high amounts of pro-inflammatory cytokines like tumour necrosis factor-alpha (TNFα) and interferon-gamma (IFNγ) that clear efficiently the pathogen3. This enhancement of the immune cells reaction after appropriate priming to stimuli totally different from the initial ones is called trained immunity and it could be a potential pathway of preventing serious infections without having severe adverse effects.

The concept has also been tested in healthy volunteers that were vaccinated with placebo or BCG (Baccillus Calmette Guérin) vaccine. These volunteers were injected 14 days latter a tri-valent influenza A vaccine. Volunteers previous vaccinated by BCG developed significantly greater titers against hemagglutinin A of the influenza A virus whereas their circulating monocytes were more potent for the production of IFNγ7. Finally, a small study has recently reported that BCG vaccination of the elderly may protect against infections8, but larger studies are necessary to confirm these findings. This generates hopes that vaccination by BCG may increase immune resistance and/or tolerance of elderly patients upon exposure to bacterial infections.

This generates hopes that vaccination by BCG may increase immune tolerance of elderly patients upon exposure to bacterial diseases.

The aim of the study is to demonstrate in a double-blind, placebo-controlled approach if vaccination of elderly patients with BCG vaccine may modulate their disease susceptibility for bacterial diseases. This will be validated using both clinical and immunological criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age more than or equal to 65 years based on the precise date of birth
* Discharge from hospital after hospitalization for a medical cause. All medical causes make patients eligible for enrolment with the only exception of medical causes mentioned in the exclusion criteria

Exclusion Criteria:

* Failure to obtain written informed consent
* Solid organ malignancy or lymphoma diagnosed the last five years
* Treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months
* Severely immunocompromised patients. This exclusion category comprises: a) patients with known infection by the human immunodeficiency virus (HIV-1); b) neutropenic patients with less than 500 neutrophils/mm3; c) patients with solid organ transplantation; d) patients with bone marrow transplantation; e) patients under chemotherapy; f) patients with primary immunodeficiency; g) severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any anti-cytokine therapies
* Positive Interferon-gamma Release Assay (IGRA)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Time to first infection | 12 months
  The time interval to the first infection post hospital discharge between the two groups of treatment.

SECONDARY OUTCOMES:
Hospitalization | Month 12
  The rate of hospitalizations will be compared between the two groups of treatment
Time to first infection or sepsis episode | Month 12
  The time to first infection or sepsis episode will be compared between the two groups of treatment
Total number of infections | Month 12
  The total number of infections will be compared between the two groups of treatment
Time to first hospitalization | Month 12
  The time to first hospitalization will be compared between the two groups of treatment
Number of antibiotic administrations | Month 12
  The number of antibiotic administrations will be compared between the two groups of treatment
Mortality | Month 12
  Mortality will be compared between the two groups of treatment
Cytokine stimulation | Month 3
  Cytokine stimulation from peripheral blood monuclear cells will be compared between the two groups of treatment
Epigenetic changes | Month 3
  Epigenetic changes of circulating monocytes will be compared between the two groups of treatment
Cost of treatment | Month 12
  The effect of BCG vaccination on cost of treatment for infections will be compared between the two groups of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Papadopoulos, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- 4th Department of Internal Medicine, ATTIKON University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leentjens J, Kox M, Stokman R, Gerretsen J, Diavatopoulos DA, van Crevel R, Rimmelzwaan GF, Pickkers P, Netea MG. BCG Vaccination Enhances the Immunogenicity of Subsequent Influenza Vaccination in Healthy Volunteers: A Randomized, Placebo-Controlled Pilot Study. J Infect Dis. 2015 Dec 15;212(12):1930-8. doi: 10.1093/infdis/jiv332. Epub 2015 Jun 12. PMID 26071565
- [Background] Blok BA, Arts RJ, van Crevel R, Benn CS, Netea MG. Trained innate immunity as underlying mechanism for the long-term, nonspecific effects of vaccines. J Leukoc Biol. 2015 Sep;98(3):347-56. doi: 10.1189/jlb.5RI0315-096R. Epub 2015 Jul 6. PMID 26150551
- [Derived] Giamarellos-Bourboulis EJ, Tsilika M, Moorlag S, Antonakos N, Kotsaki A, Dominguez-Andres J, Kyriazopoulou E, Gkavogianni T, Adami ME, Damoraki G, Koufargyris P, Karageorgos A, Bolanou A, Koenen H, van Crevel R, Droggiti DI, Renieris G, Papadopoulos A, Netea MG. Activate: Randomized Clinical Trial of BCG Vaccination against Infection in the Elderly. Cell. 2020 Oct 15;183(2):315-323.e9. doi: 10.1016/j.cell.2020.08.051. Epub 2020 Sep 1. PMID 32941801